CLINICAL TRIAL: NCT04130776
Title: Demonstrating the Stability of the Analytes Measured for 4Kscore: Total PSA (tPSA), Free PSA (fPSA), Intact PSA (iPSA), and Human Kallikrein 2 (hk2) in Clinical Serum Samples Stored Uncentrifuged Before Testing
Brief Title: 4Kscore Using Serum Stored Uncentrifuged
Status: Completed | Type: Observational
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 20622
Record Dates: First submitted 2019-10-10; First posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Measurement of four prostate-specific kallikreins for the 4Kscore Test when serum stored uncentrifuged — The 4Kscore Test helps clarify the biopsy decision-making process by determining a patient specific probability for finding aggressive, Gleason score 7 or higher prostate cancer upon biopsy. These are the aggressive prostate cancers that always require medical treatment or intervention. The 4Kscore Test relies on the measurement of four prostate-specific kallikreins in the blood: Total PSA, Free PSA, Intact PSA, and Human Kallikrein 2 (hK2). The blood test results are combined in an algorithm with patient age, digital rectal exam (nodules, no nodules), and prior negative biopsy (yes, no) to give physicians a personal score for each patient. The 4Kscore Test predicts the risk percent score from <1% to >95% of a man having aggressive cancer in a prospective biopsy.

SUMMARY:
The purpose of the study is to evaluate whether storage of serum uncentrifuged is an allowable preanalytical procedure

ELIGIBILITY:
Inclusion Criteria:

* Men capable of donating five 5 mL tubes of whole blood
* 40 to 80 years old
* No prior diagnosis of prostate cancer; prior negative prostate biopsy included
* Total PSA (tPSA) value measured within last year to be: at 1.5 ng/mL to 4 ng/mL, 4.1 ng/mL to 10 ng/mL and 10 ng/mL and above

Exclusion Criteria:

* In the previous 96 hours (4 days), underwent a digital rectal exam
* Any invasive urologic procedure in the 6 months prior to study participation
* Underwent any procedure to treat symptomatic benign prostatic hyperplasia in the last 6 months
* Radical prostatectomy since tPSA measurement
* Received within the previous 6 months 5-alpha reductase inhibitor (5-ARI) therapy such as Avodart (dutasteride) or Proscar (finasteride)

Ages: 40 Years to 80 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: The study population will be 40 to 80 years old male whom have met all eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2018-03-27 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
tPSA changes in 3 days | Day 0, 1, 2 and 3
  Measure tPSA in serum samples at day 0, 1, 2 and 3
fPSA changes in 3 days | Day 0, 1, 2 and 3
  Measure fPSA in serum samples at day 0, 1, 2 and 3
iPSA changes in 3 days | Day 0, 1, 2 and 3
  Measure iPSA in serum samples at day 0, 1, 2 and 3
hK2 changes in 3 days | Day 0, 1, 2 and 3
  Measure hK2 in serum samples at day 0, 1, 2 and 3

CONTACTS AND LOCATIONS:
Overall Officials: James Ryan Mark, Principal Investigator — Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States